CLINICAL TRIAL: NCT07360067
Title: Prospective Cohort Study of Bachmann Bundle Versus Right Atrial Appendage Pacing: Impact on Atrial Cardiomyopathy Evaluated by Echocardiographic Parameters and Clinical Outcome
Acronym: BRAVE
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC2025-10-106; KCT0011382 (Other: Korea National Institute of Health)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sick Sinus Syndrome
Keywords: bachmann bundle pacing
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Right Atrial Appendage Pacing: Right Atrial Appendage Pacing
  Interventions: Procedure: Right Atrial Appendage Pacing
- Bachmann Bundle Pacing: Bachmann Bundle Pacing
  Interventions: Procedure: Bachmann Bundle Pacing

INTERVENTIONS:
Procedure: Right Atrial Appendage Pacing — Atrial lead positioned in the right atrial appendage
  Groups: Right Atrial Appendage Pacing
Procedure: Bachmann Bundle Pacing — Atrial lead positioned in the bachmann bundle branch
  Groups: Bachmann Bundle Pacing

SUMMARY:
The goal of this observational study is to evaluate the impact of different atrial pacing sites-Bachmann's bundle pacing versus right atrial appendage pacing-on the development and progression of atrial cardiomyopathy in patients diagnosed with sick sinus syndrome who are undergoing permanent pacemaker implantation.

DETAILED DESCRIPTION:
Previous studies have reported that conventional Right Atrial Appendage pacing is associated with delayed atrial activation time. A higher burden of atrial pacing at this site has been linked to an increased incidence of atrial fibrillation and atrial tachycardia. Furthermore, structural and functional deterioration of the atria-specifically Left Atrial dilation and reduced left atrial strain-has been observed in patients with a high percentage of Right Atrial Appendage pacing. These changes are known to accelerate the progression of atrial cardiomyopathy, potentially leading to adverse long-term clinical outcomes.

To address these limitations, Bachmann Bundle Pacing has emerged as a promising alternative pacing site. The Bachmann bundle is a major atrial myoarchitecture connecting the right and left atria. Pacing at this site is expected to facilitate interatrial conduction, thereby restoring interatrial synchrony and mitigating interatrial block. Prior research indicates that pacing at the Bachmann bundle is associated with a reduced incidence of atrial fibrillation and atrial tachycardia, suggesting distinct benefits regarding atrial electrophysiological outcomes. However, existing studies have primarily focused on electrophysiological parameters, such as arrhythmia incidence. Consequently, the impact of Bachmann Bundle Pacing on atrial structural and functional remodeling remains to be clearly elucidated.

Therefore, this study is designed as a single-center cohort study enrolling a total of 200 subjects (100 prospective and 100 retrospective). We will analyze echocardiographic parameters over a 12-month period following pacemaker implantation. By comprehensively analyzing imaging parameters (left atrial/right atrial strain and volume changes assessed via echocardiography) and clinical outcomes (atrial arrhythmias, heart failure hospitalization, and mortality), this study aims to investigate the differential effects of Bachmann Bundle Pacing versus Right Atrial Appendage pacing on the development and progression of atrial cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older
* Patients diagnosed with sick sinus syndrome who are scheduled for de novo implantation of a permanent pacemaker or permanent implantable cardioverter-defibrillator
* Patients or their legal representatives who voluntarily consent to the access of medical records and study data throughout the entire research period

Exclusion Criteria:

* Patients with persistent or permanent AF
* Patients with a life expectancy of less than one year due to other comorbidities
* Pregnant or breastfeeding women
* Patients who refuse active treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to Samsung Medical Center, were diagnosed with Sick Sinus Syndrome, and underwent de novo permanent pacemaker or implantable cardioverter-defibrillator implantation based on clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural echocardiographic parameters of the left atrium | 6 and 12 months after pacemaker implantation
  LA Volume Index measured as mL/m^2
Functional echocardiographic parameters of the left atrium | 6 and 12 months after pacemaker implantation
  Reservoir Strain (%), Conduit Strain (%), Contraction Strain (%)

SECONDARY OUTCOMES:
Structural echocardiographic parameters of the left ventricle | 6 and 12 months after pacemaker implantation
  LV End-Diastolic Diameter(mm), LV End-Systolic Diameter(mm)
Functional echocardiographic parameters of the left ventricle | 6 and 12 months after pacemaker implantation
  LV Ejection Fraction (%), Global Longitudinal Strain (%)
Mitral and tricuspid regurgitation volume | 6 and 12 months after pacemaker implantation
  as mL per beat
Structural echocardiographic parameters of the right atrium | 6 and 12 months after pacemaker implantation
  RA Volume Index (mL/m^2)
Functional echocardiographic parameters of the right atrium | 6 and 12 months after pacemaker implantation
  RA Reservoir Strain (%), RA Conduit Strain (%), RA Contraction Strain (%)
ECG parameters | 6 and 12 months after pacemaker implantation
  PR interval (ms), QRS duration (ms), P wave duration (ms), QTC (ms)
Average heart rate | 6 and 12 months after pacemaker implantation
  bpm
Heart rate distribution | 6 and 12 months after pacemaker implantation
  percentage (%)
Pacing burden | 6 and 12 months after pacemaker implantation
  percentage (%)
Atrial fibrillation burden | 6 and 12 months after pacemaker implantation
  percentage (%)
atrial fibrillation occurrence | 6 and 12 months after pacemaker implantation
  count
NTproBNP | 6 and 12 months after pacemaker implantation
  pg/ml
Procedure-related complications | 6 and 12 months after pacemaker implantation
  count
Pacemaker/Implantable cardioverter defibrillator parameters | 6 and 12 months after pacemaker implantation
  Threshold (V)
Pacemaker/Implantable cardioverter defibrillator parameters | 6 and 12 months after pacemaker implantation
  longevity (year)
Cardiac mortality | 6 and 12 months after pacemaker implantation
  count
All-cause mortality | 6 and 12 months after pacemaker implantation
  count
Patient's functional status | 6 and 12 months after pacemaker implantation
  NYHA class I~IV
hospitalization due to heart failure | 6 and 12 months post-procedure
  count
re-admission due to any cause | 6 and 12 months post-procedure
  count
Cerebrovascular event | 6 and 12 months post-procedure
  count

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bailin SJ, Adler S, Giudici M. Prevention of chronic atrial fibrillation by pacing in the region of Bachmann's bundle: results of a multicenter randomized trial. J Cardiovasc Electrophysiol. 2001 Aug;12(8):912-7. doi: 10.1046/j.1540-8167.2001.00912.x. PMID 11513442
- [Result] Infeld M, Nicoli CD, Meagher S, Tompkins BJ, Wayne S, Irvine B, Betageri O, Habel N, Till S, Lobel J, Meyer M, Lustgarten DL. Clinical impact of Bachmann's bundle pacing defined by electrocardiographic criteria on atrial arrhythmia outcomes. Europace. 2022 Oct 13;24(9):1460-1468. doi: 10.1093/europace/euac029. PMID 35304608
- [Result] Lustgarten DL, Habel N, Sanchez-Quintana D, Winget J, Correa de Sa D, Lobel R, Thompson N, Infeld M, Meyer M. Bachmann bundle pacing. Heart Rhythm. 2024 Sep;21(9):1711-1717. doi: 10.1016/j.hrthm.2024.03.1786. Epub 2024 Mar 27. No abstract available. PMID 38552731
- [Result] Martens P, Deferm S, Bertrand PB, Verbrugge FH, Ramaekers J, Verhaert D, Dupont M, Vandervoort PM, Mullens W. The Detrimental Effect of RA Pacing on LA Function and Clinical Outcome in Cardiac Resynchronization Therapy. JACC Cardiovasc Imaging. 2020 Apr;13(4):895-906. doi: 10.1016/j.jcmg.2019.04.022. Epub 2019 Jul 17. PMID 31326478
- [Result] Roithinger FX, Abou-Harb M, Pachinger O, Hintringer F. The effect of the atrial pacing site on the total atrial activation time. Pacing Clin Electrophysiol. 2001 Mar;24(3):316-22. doi: 10.1046/j.1460-9592.2001.00316.x. PMID 11310300
- [Result] De Sisti A, Leclercq JF, Stiubei M, Fiorello P, Halimi F, Attuel P. P wave duration and morphology predict atrial fibrillation recurrence in patients with sinus node dysfunction and atrial-based pacemaker. Pacing Clin Electrophysiol. 2002 Nov;25(11):1546-54. doi: 10.1046/j.1460-9592.2002.01546.x. PMID 12494610
- [Result] Elkayam LU, Koehler JL, Sheldon TJ, Glotzer TV, Rosenthal LS, Lamas GA. The influence of atrial and ventricular pacing on the incidence of atrial fibrillation: a meta-analysis. Pacing Clin Electrophysiol. 2011 Dec;34(12):1593-9. doi: 10.1111/j.1540-8159.2011.03192.x. Epub 2011 Aug 7. PMID 21819434
- [Result] Bradshaw PJ, Stobie P, Knuiman MW, Briffa TG, Hobbs MS. Trends in the incidence and prevalence of cardiac pacemaker insertions in an ageing population. Open Heart. 2014 Dec 10;1(1):e000177. doi: 10.1136/openhrt-2014-000177. eCollection 2014. PMID 25512875
- [Result] Honarbakhsh S, Hunter L, Chow A, Hunter RJ. Bradyarrhythmias and pacemakers. BMJ. 2018 Mar 15;360:k642. doi: 10.1136/bmj.k642. No abstract available. PMID 29545242
- [Result] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2019 Aug 20;140(8):e382-e482. doi: 10.1161/CIR.0000000000000628. Epub 2018 Nov 6. No abstract available. PMID 30586772